CLINICAL TRIAL: NCT01451203
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of CDP870 in Patients With Early-stage Rheumatoid Arthritis Who Are Naïve to Methotrexate and Have Poor Prognostic Factors
Brief Title: Efficacy Confirmation Study of CDP870 in Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDP870-275-11-001; JapicCTI-111636 (Other: JAPIC)
Record Dates: First submitted 2011-09-25; First posted 2011-10-13 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Cimzia; Early RA; Certolizumab Pegol
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBO + MTX (Placebo Comparator): Participants who received placebo subcutaneously every two weeks (Q2W) at Weeks 0, 2, and 4; followed by placebo subcutaneously Q2W from Week 6 to Week 50 and an oral dose of MTX administered from Week 0 onwards
  Interventions: Drug: Placebo; Drug: methotrexate (MTX)
- CZP + MTX (Experimental): Participants who certolizumab pegol (CZP) subcutaneously at a loading dose of CZP 400 mg every 2 weeks (Q2W) at Weeks 0, 2, and 4; followed by a dose of CZP 200 mg subcutaneously Q2W from Week 6 to Week 50 and an oral dose of MTX administered from Week 0 onwards
  Interventions: Drug: CZP; Drug: methotrexate (MTX)

INTERVENTIONS:
Drug: Placebo — Subcutaneous (SC)
  Arms: PBO + MTX
Drug: CZP — SC
  Other Names: CDP870; certolizumab pegol; Cimzia®
  Arms: CZP + MTX
Drug: methotrexate (MTX) — oral

SUMMARY:
The objective of this study is to assess the efficacy of certolizumab pegol (CZP) with methotrexate (MTX) compared with MTX-alone in patients with early-stage rheumatoid arthritis (RA) who are naive to MTX and have with poor prognostic factors, using inhibition of radiographically confirmed joint damage progression over a one-year period as a primary endpoint. Following a year of treatment with CZP plus MTX treatment, CZP will be discontinued, and the subjects will be monitored for one more year (the follow-up period) to investigate the sustainability of efficacy of CZP during the MTX monotherapy for exploratory purposes.

DETAILED DESCRIPTION:
This study was initiated by Otsuka Pharmaceutical Co., Ltd and transferred to Astellas on 12/04/2012.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with RA as defined by the ACR/EULAR criteria (2010) who meet all of the following criteria:

  1. Subjects who developed RA within one year after onset of RA.
  2. Subjects who have never received MTX before (MTX naive)
  3. Subjects whose disease activity is moderate or higher (DAS28(ESR) ≥ 3.2）
  4. Subjects must satisfy at least two of the three criteria (Anti-CCP antibody positive, Rheumatoid factor positive, Presence of X-ray erosion） for poor prognostic factors. The anti-CCP antibody positive is essential for every patient.

Exclusion Criteria:

* Patients who have a diagnosis of any other type of inflammatory arthritis.
* Patients who have a secondary, non-inflammatory type of arthritis.
* Patients who have used with MTX, reflunomide, or any other biologics prior to the start of study drug administration.
* Patients who have NYHA (New York Heart Association) Class III or IV congestive heart failure
* Patients who currently have, or who have a history of, tuberculosis.
* Patients who have a high risk of infection (with a current infectious disease, a chronic infectious disease, a history of serious infectious disease)
* Patients who currently have, or have a history of, malignant tumor
* Female patients who are breastfeeding or pregnant, who are of childbearing potential

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 319 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2013-08-28 (Actual); Study Completion 2014-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Atsumi T, Tanaka Y, Yamamoto K, Takeuchi T, Yamanaka H, Ishiguro N, Eguchi K, Watanabe A, Origasa H, Yasuda S, Yamanishi Y, Kita Y, Matsubara T, Iwamoto M, Shoji T, Togo O, Okada T, van der Heijde D, Miyasaka N, Koike T. Clinical benefit of 1-year certolizumab pegol (CZP) add-on therapy to methotrexate treatment in patients with early rheumatoid arthritis was observed following CZP discontinuation: 2-year results of the C-OPERA study, a phase III randomised trial. Ann Rheum Dis. 2017 Aug;76(8):1348-1356. doi: 10.1136/annrheumdis-2016-210246. Epub 2017 Feb 2. PMID 28153828
- [Derived] Atsumi T, Yamamoto K, Takeuchi T, Yamanaka H, Ishiguro N, Tanaka Y, Eguchi K, Watanabe A, Origasa H, Yasuda S, Yamanishi Y, Kita Y, Matsubara T, Iwamoto M, Shoji T, Okada T, van der Heijde D, Miyasaka N, Koike T. The first double-blind, randomised, parallel-group certolizumab pegol study in methotrexate-naive early rheumatoid arthritis patients with poor prognostic factors, C-OPERA, shows inhibition of radiographic progression. Ann Rheum Dis. 2016 Jan;75(1):75-83. doi: 10.1136/annrheumdis-2015-207511. Epub 2015 Jul 2. PMID 26139005
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=CDP870-275-11-001/1226-CL-B001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with early rheumatoid arthritis (RA), methotrexate (MTX)-naïve and had poor prognostic factors were recruited for this study.
Groups:
- CZP + MTX: Participants who received certolizumab pegol (CZP) subcutaneously at a loading dose of CZP 400 mg every 2 weeks (Q2W) at Weeks 0, 2, and 4; followed by a dose of CZP 200 mg subcutaneously Q2W from Week 6 to Week 50 and an oral dose of MTX administered from Week 0 onwards
Period: Double-blind Treatment Period
Arm/Group | PBO + MTX | CZP + MTX
Started | 158 | 161
Received Treatment | 157 | 159
Received Rescue Treatment | 70 (Participants who did not achieve improvement at & after Week 24 were dropped out of study schedule.) | 36 (Participants who did not achieve improvement at & after Week 24 were dropped out of study schedule.)
Completed | 73 | 111
Not Completed | 85 | 50
Not completed — Did not receive treatment | 1 | 2
Not completed — Consent Withdrawn | 3 | 2
Not completed — Lack of Efficacy | 71 | 36
Not completed — HBV-DNA positive (during the DB Period) | 0 | 1
Not completed — Adverse Event | 6 | 9
Not completed — Missing study medication ≥6 times | 1 | 0
Not completed — Violation of eligibility criteria | 1 | 0
Not completed — Investigator decision | 2 | 0
Period: Post-treatment Period
Arm/Group | PBO + MTX | CZP + MTX
Started | 71 (Two participants received rescue treatment and did not enter this period.) | 108 (Three participants received rescue treatment and did not enter this period.)
Received Rescue Treatment | 12 (Participants who presented with flares at any time were dropped out of study schedule.) | 28 (Participants who presented with flares at any time were dropped out of study schedule.)
Completed | 57 | 74
Not Completed | 14 | 34
Not completed — Consent withdrawn | 2 | 4
Not completed — Lack of Efficacy | 12 | 28
Not completed — Adverse Event | 0 | 1
Not completed — Investigator decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS), which consisted of all participants who had received at least 1 study drug administration and provided efficacy data after the administration of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PBO + MTX | CZP + MTX | Total
Number analyzed (Participants) | 157 | 159 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (10.3) | 49.4 (10.6) | 49.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 129 | 256
  Male | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 52
Description: Radiographs/X-rays of hands and feet (posteroanterior views of both hands and dorsoplantar views of both feet) were independently assessed by two radiographic readers. The degree of joint damage was graded by assessing bone erosion in 44 joints and joint space narrowing (JSN) in 42 joints. The bone erosion score is a summary of erosion severity in 32 joints of the hands and 12 joints in the feet. Each joint was scored, according to the surface area involved, from 0 (no erosion) to 5 (complete collapse of bone). The score for erosion ranges from 0 to 160 in the hands and from 0 to 120 in the feet (the maximum erosion score for a joint in the foot is 10). The JSN score summarizes the severity of JSN in 30 joints of the hands and 12 joints of the feet. JSN, including subluxation, was scored from 0 (normal) to 4 (complete loss of joint space, bony ankylosis, or luxation), with a maximum JSN score of 168. The mTSS ranges from 0 (normal) to 448 (worst).
Time Frame: Baseline and Week 52
Population: FAS with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PBO + MTX | CZP + MTX
Number analyzed (Participants) | 157 | 158
units on a scale | 1.58 (4.86) | 0.36 (2.70)
Statistical Analysis 1: Comparison: PBO + MTX vs CZP + MTX; The mTSS was analyzed using LINEAR for the imputation of missing data at Week 52.The primary Week 52 analysis assessed whether treatment up to Week 52 with the CZP group was superior to the placebo group in mTSS at Week 52. The 2-sided null and alternative hypotheses were: H0: πC = πM Ha: πC ≠ πM where πC represented subjects in the CZP group at Week 52 and πM represented subjects in the placebo group at Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA — The ANCOVA on the ranks with treatment as factors and Baseline rank as covariate was used; Hodges-Lehmann point estimate of shift = 0.00, 95% CI 2-sided [0.00 to 0.00]

2. Secondary Outcome: Change From Baseline in mTSS at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: FAS with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PBO + MTX | CZP + MTX
Number analyzed (Participants) | 157 | 158
units on a scale | 0.86 (2.37) | 0.26 (1.55)
Statistical Analysis 1: Comparison: PBO + MTX vs CZP + MTX; The mTSS was analyzed using LINEAR for the imputation of missing data at Week 24; Test type: Superiority or Other; p = 0.003, ANCOVA; The ANCOVA on the ranks with treatment as factors and Baseline rank as covariate was used; Hodges-Lehman point estimate of shift = 0.00, 95% CI 2-sided [0.00 to 0.00]

3. Secondary Outcome: Clinical Remission Rate: Percentage of Participants Meeting the Disease Activity Score-28 Joint Count (DAS28) Erythrocyte Sedimentation Rate (ESR) (DAS28[ESR]) Remission Criteria at Weeks 24 and 52
Description: The DAS28(ESR) measures the severity of disease at a specific time and is derived from the following variables: •28 tender joint count (TJC); •28 swollen joint count (SJC); •ESR; •Patient's global assessment of disease activity (PtGADA). To obtain the tender joint count and swollen joint count, 28 joints of the shoulder, elbow, wrist, metacarpophalangeal joints, thumb interphalangeal joints, proximal interphalangeal joints, and knee joints were examined. DAS28(ESR) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible ESR. A participant was considered to be in remission if DAS28(ESR) <2.6. Last Observation Carried Forward" (LOCF) was applied.
Time Frame: Week 24 and Week 52
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBO + MTX | CZP + MTX
Number analyzed (Participants) | 157 | 159
percentage of participants
  Week 24 | 30.6 [23.5 to 38.4] | 52.8 [44.8 to 60.8]
  Week 52 | 36.9 [29.4 to 45.0] | 57.2 [49.2 to 65.0]
Statistical Analysis 1: Comparison: PBO + MTX vs CZP + MTX; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Secondary Outcome: Clinical Remission Rate: Percentage of Participants Meeting the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Simplified Disease Activity Index (SDAI)-Based Remission Criteria at Weeks 24 and 52
Description: The ACR/EULAR SDAI remission rate measures the severity of disease at a specific time and is derived from the following variables: •28 tender joint count (TJC); •28 swollen joint count (SJC); •Patient's global assessment of disease activity (PtGADA); •Physician's Global Assessment of Disease Activity (PhGADA); •C-reactive protein (CRP) To obtain the tender joint count and swollen joint count, 28 joints of the shoulder, elbow, wrist, metacarpophalangeal joints, thumb interphalangeal joints, proximal interphalangeal joints, and knee joints were examined. A participant was considered to be in remission if SDAI ≤3.3. Last Observation Carried Forward (LOCF) was applied.
Time Frame: Week 24 and Week 52
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBO + MTX | CZP + MTX
Number analyzed (Participants) | 157 | 159
percentage of participants
  Week 24 | 29.3 [22.3 to 37.1] | 48.4 [40.4 to 56.5]
  Week 52 | 33.8 [26.4 to 41.7] | 57.9 [49.8 to 65.6]
Statistical Analysis 1: Comparison: PBO + MTX vs CZP + MTX; Test type: Superiority or Other; p < 0.001, Fisher Exact

5. Secondary Outcome: Percentage of Participants Meeting the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Boolean-based Remission Criteria at Weeks 24 and 52
Description: The ACR/EULAR Boolean-based remission rate measures the severity of disease at a specific time and is derived from the following variables: •28 tender joint count (TJC); •28 swollen joint count (SJC); •Patient's global assessment of disease activity (PtGADA); •C-reactive protein (CRP) To obtain the tender joint count and swollen joint count, 28 joints of the shoulder, elbow, wrist, metacarpophalangeal joints, thumb interphalangeal joints, proximal interphalangeal joints, and knee joints were examined. A participant was considered to be in remission if all the criteria for each variable was met:TJC (in 28 joints) ≤1; SJC (in 28 joints) ≤1; CRP ≤1 mg/dl; PtGADA ≤1. Last Observation Carried Forward (LOCF) was applied
Time Frame: Week 24 and Week 52
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBO + MTX | CZP + MTX
Number analyzed (Participants) | 157 | 159
percentage of participants
  Week 24 | 22.3 [16.0 to 29.6] | 36.5 [29.0 to 44.5]
  Week 52 | 28.0 [21.2 to 35.7] | 45.3 [37.4 to 53.4]
Statistical Analysis 1: Comparison: PBO + MTX vs CZP + MTX; Test type: Superiority or Other; p = 0.002, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to last dose of study drug (up to 104 weeks)
Arm/Group | PBO + MTX | CZP + MTX
Serious Adverse Events (participants affected / at risk) | 18/157 | 17/159
Other Adverse Events (participants affected / at risk) | 139/157 | 146/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBO + MTX (N=157) | CZP + MTX (N=159)
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 | 3
Bronchitis (Infections and infestations) | 0 | 1
Meningitis fungal (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Crush injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PBO + MTX (N=157) | CZP + MTX (N=159)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 9
Nausea (Gastrointestinal disorders) | 30 | 39
Stomatitis (Gastrointestinal disorders) | 27 | 27
Abdominal discomfort (Gastrointestinal disorders) | 9 | 16
Dental caries (Gastrointestinal disorders) | 10 | 14
Constipation (Gastrointestinal disorders) | 3 | 10
Abdominal pain upper (Gastrointestinal disorders) | 3 | 9
Vomiting (Gastrointestinal disorders) | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 10 | 6
Gastritis (Gastrointestinal disorders) | 10 | 4
Malaise (General disorders) | 11 | 14
Hepatic function abnormal (Hepatobiliary disorders) | 48 | 51
Liver disorder (Hepatobiliary disorders) | 9 | 9
Nasopharyngitis (Infections and infestations) | 54 | 70
Pharyngitis (Infections and infestations) | 13 | 24
Gastroenteritis (Infections and infestations) | 10 | 19
Bronchitis (Infections and infestations) | 13 | 12
Upper respiratory tract infection (Infections and infestations) | 11 | 10
Oral herpes (Infections and infestations) | 8 | 6
White blood cell count decreased (Investigations) | 7 | 10
Cell marker increased (Investigations) | 1 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 3
Headache (Nervous system disorders) | 8 | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Eczema (Skin and subcutaneous tissue disorders) | 7 | 13
Rash (Skin and subcutaneous tissue disorders) | 3 | 13

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for to seek patent protection.